CLINICAL TRIAL: NCT07012915
Title: Immunological-Clinical Evaluation of the Etiopathogenesis of Peri-Implantitis
Acronym: PERI-EDU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Collaborators: University of Bern (Other); University of Barcelona (Other); University of Roma La Sapienza (Other); Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KA220-HED
Record Dates: First submitted 2025-05-14; First posted 2025-06-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-05

CONDITIONS: Peri-Implantitis
Keywords: Perii-implantitis; Titanium alloys corosion; Titanium implants
MeSH Terms: conditions — Peri-Implantitis | interventions — Hematologic Tests; Radiation

STUDY DESIGN:
Intervention Model Description: Healthy adult participants, suffering from Peri-Implantitis. Every participant from a total number of 100 will have blood sample collected twice before and 4 weeks following implant removal for detailed evaluation. Furthermore, the Cone Beam Computed Tomography will be applied to evaluate the severity and shape of bone defect. Removed implants will be send for detailed chemical evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Every participant will achieve same intervention when it comes to surgical treatment, clinical examination, radiology evaluation and defined parameters of blood serum.
  Interventions: Diagnostic Test: Blood testing

INTERVENTIONS:
Diagnostic Test: Blood testing — Blood sample will be collected twice for each participants procedding and following dental implant removal. Cone Beam Computed Tomography will be applied to evaluate the shape, severity of bone defect in direct viscinity of the implant.
  Other Names: Radiation; Surgery

SUMMARY:
A total of 100 adult volunteers of both sexes will be enrolled in the project. The study will be conducted within an international consortium formed for the project, comprising the following institutions: Wroclaw Medical University (Poland), Sapienza University of Rome (Italy), University of Barcelona (Spain), University of Bern (Switzerland), and Egas Moniz University (Portugal). Each international partner institution will recruit 20 volunteers as participants in the experiment. Each of the participating institutions will submit an application to their respective local bioethics committee for approval to conduct the medical experiment. Each partner institution will conduct procedures at their respective clinical locations.

Eligibility Criteria participants must have undergone previous implant treatment that has resulted in active, advanced peri-implantitis. Exclusion Criteria: General and local contraindications for surgical procedures Pregnancy; Use of bisphosphonates or other antiresorptive medications in medical history Laboratory Analysis Procedures.

During the initial visit, patients will undergo a medical interview and a dental examination with regard to: Oral Hygiene Indices; Periodontal disease indices. For the implant site, the following parameters will be evaluated: Pocket Depth Bleeding on Probing Width and height of the attached gingiva Possible implant mobility, assessed using the Mobility Index Following the clinical examination, each participant will be referred for a Cone Beam Computed Tomography (CBCT) scan with measurements including: Bone loss percentage for each of the four implant surfaces, Bone density. Next, a 20ml venous blood sample will be collected from the antecubital vein of each participant and sent to a laboratory for further analysis, including: Hematological Inflammation Indices: Systemic Immune-Inflammation Index, Aggregate Index of Systemic Inflammation, Complete blood count, Lipid profile, APOA., APOBg, Inflammatory markers, albumin, total protein, total ferritin, fibrinogen, Cytokine profile, HOMA2 Parameters, Thyroid profile, Vitamin D level Next, each participant will undergo implant explantation surgery, during which tissue samples will be collected for further analysis. Implant surface will be analyzed using: light microscopy, scanning electron microscopy, corrosion testing.

Follow-Up will be scheduled four weeks later with following evaluation: Clinical assessment of the implantation site. A CBCT scan to assess bone structure in the post-implantation region, with measurements including percentage of bone loss. Moreover, 20ml of venous blood will be collected from the antecubital vein of each participant. The blood sample will be preserved and sent to an analytical laboratory for further testing, including for same as previously mentioned tests.

DETAILED DESCRIPTION:
The following research experiment project is part of the scientific section of a project funded under the Erasmus+ program (KA220-HED - Cooperation partnerships in higher education) entitled "Integrating Peri-Implantitis Research into Higher Education Curriculum - Developing and Integrating Evidence-Based Teaching Materials and Clinical Tools." According to the current state of knowledge, there are two main theories explaining the development of peri-implantitis. The first theory suggests that the primary etiological factor is the invasion of periopathogens along the gingival crevice surrounding the implant, resembling the pathogenic development seen in natural periodontal diseases such as gingivitis and periodontitis. In this scenario, bacterial invasion is facilitated by the distinct structure of the peri-implant soft tissues, which differ from natural gingival tissue in several ways: a more uniaxial, parallel orientation of collagen fibers relative to the implant's long axis, lower cellular density, and reduced mitotic potential of the surrounding soft tissue.

The second theory proposes that marginal bone loss around the implant is the result of an immuno-osteolytic reaction, with pathogenic bacteria appearing as a secondary phenomenon. According to this theory, the initiation of the pathological process is attributed to an immune response triggered by the presence of titanium ions and other metallic elements, such as vanadium, which is commonly found in titanium alloys. In vitro models have demonstrated that an increase in Ti concentration leads to macrophage activation and increased secretion of pro-inflammatory cytokines, particularly interleukin IL-1B and arachidonic acid derivatives. This macrophage activation is significantly higher in cases where prior bacterial lipopolysaccharide (LPS) exposure has occurred, suggesting an additive effect of bacterial factors in the overall disease process. Furthermore, vanadium appears to disrupt the balance of T/B lymphocytes, suppress the secretion of anti-inflammatory cytokines, and activate the innate immune response via Toll-like receptors and NF-κB signaling pathways.

Despite conceptual differences between these two theories, both agree on the fundamental premise that biological processes occurring on the implant surface and in its immediate vicinity play a critical role in the development of peri-implantitis. These processes are modulated by the physicochemical properties of the implant surface.

The immuno-osteolytic concept of peri-implantitis, also known as the foreign body reaction theory, is largely based on physicochemical changes that occur on the implant surface over time due to its exposure to the oral tissue environment. These changes are associated with gradual degradation, corrosion, and aging of titanium alloys.

In biomedical applications, biphasic titanium alloys are most commonly used, particularly the Ti-6Al-4V alloy, which contains 6% aluminum and 4% vanadium. Aluminum stabilizes the α-phase, improving mechanical strength and reducing weight, while vanadium stabilizes the β-phase, enhancing alloy plasticity.

All known metals and alloys undergo corrosion under specific conditions. Most of them are thermodynamically unstable, tending to transition from their metallic state to ionic form. The degree of thermodynamic stability of a metal is characterized by its standard electrode potential, which describes the free energy change when an ion transitions from the metal to a solution. The more negative the standard electrode potential, the lower the metal's resistance to corrosion. The standard ionization potential of titanium is theoretically established at 1.63V, indicating high electrochemical potential and corrosion susceptibility of pure titanium. However, in practice, titanium exhibits lower corrosion potential due to its tendency to undergo passivation, forming a stable oxide layer that acts as a barrier preventing direct contact between the metal and the external environment.

The stability of the titanium dioxide (TiO₂) passive layer in the oral cavity is compromised by salivary enzymes and bacterial metabolism, particularly acidic byproducts such as lactic, acetic, and propionic acids. These substances create localized pH shifts towards acidity, which are unfavorable for titanium alloys and accelerate corrosion. Another factor increasing titanium corrosion in dental applications is the presence of fluoride compounds, which are commonly used in toothpaste, mouthwashes, gels, and fluoride foams. In aqueous solutions, fluoride exists primarily as the fluoride ion (F-), which has the ability to dissolve the passive oxide layer on titanium, significantly increasing corrosion rates.

A separate concern is the fatigue-related degradation of titanium implants. These fatigue processes are associated with repeated mechanical stress, particularly non-linear loading patterns. The first observable sign of fatigue is the formation of microcracks, detectable via scanning electron microscopy (SEM). In advanced stages, these microcracks lead to wear-corrosion phenomena, further accelerating surface degradation of titanium alloys.

Objectives of the Medical Experiment:

Clinical assessment of oral health, with a particular focus on periodontal indicators and oral hygiene status in participants affected by peri-implantitis.

Radiological evaluation of bone structure affected by peri-implantitis. Hematological assessment of peri-implantitis markers and the immunological profile of participants diagnosed with peri-implantitis.

Measurement of Ti++ ion concentrations and other metallic elements present in titanium alloys in tissues surrounding implants affected by peri-implantitis.

Corrosion analysis and SEM-based fatigue analysis of implant surfaces associated with peri-implantitis.

Study design A total of 100 adult volunteers of both sexes will be enrolled in the project. The study will be conducted within an international consortium formed for the project, comprising the following institutions: Wroclaw Medical University (Poland), Sapienza University of Rome (Italy), University of Barcelona (Spain), University of Bern (Switzerland), and Egas Moniz University (Portugal).

Each international partner institution will recruit 20 volunteers as participants in the experiment. Each of the participating institutions (Sapienza University of Rome, University of Barcelona, University of Bern, and Egas Moniz University) will submit an application to their respective local bioethics committee for approval to conduct the medical experiment.

Eligibility Criteria To be eligible for the study, participants must have undergone previous implant treatment that has resulted in active, advanced peri-implantitis.

During the initial visit, patients will undergo a medical interview to document their systemic diseases and dental treatment history, with particular emphasis on:

The type and brand of implant The prosthetic loading type of the implant The location and time of implantation The onset and treatment history of peri-implantitis

Each participant will then undergo a dental examination, utilizing a UNC15 periodontal probe (DepplerSA, Roller, Switzerland). This assessment will include:

Oral hygiene indicators: Oral Hygiene Index (OHI), Aproximal Plaque Index (API) Periodontal disease indices: Community Index of Periodontal Treatment Needs (CPITN) Occlusal abnormalities and increased facial muscle tension, particularly in the mentalis muscle and oral floor muscles Implant-Specific Assessments

For the implant site, the following parameters will be evaluated:

Pocket Depth (PD) - measured on four surfaces around the implant Bleeding on Probing (BoP) Index Width and height of the attached gingiva (HKT, WKT) Possible implant mobility, assessed using the Mobility Index (MOB) Following the clinical examination, each participant will be referred for a Cone Beam Computed Tomography (CBCT) scan.

CBCT Examination

The CBCT scan will be routinely evaluated, focusing on the implant region, with measurements including:

Bone loss percentage, calculated as the ratio of bone defect depth from the implant platform to the base of the defect, relative to the total implant length, assessed separately for each of the four implant surfaces (mesial, distal, buccal, and lingual/palatal).

Bone density, measured in Hounsfield units (HU)

A peri-implantitis process will be classified as active if:

PD at the implant site exceeds 6mm, with a positive BoP index Advanced peri-implantitis is diagnosed if bone loss exceeds 66% on at least one implant surface Treatment Eligibility Criteria According to established literature, in cases of active, advanced peri-implantitis, where bone loss exceeds 50% of the implant length, implant removal is considered the appropriate therapeutic approach. Only patients meeting this criterion will be enrolled in the project.

Exclusion Criteria:

General and local contraindications for surgical procedures Pregnancy Use of bisphosphonates or other antiresorptive medications in medical history Patients who do not meet the implant removal criteria and are not eligible for the study will be directed toward non-surgical or conservative-surgical treatment options.

Laboratory Analysis Procedures

During a subsequent procedural visit, a 20ml venous blood sample will be collected from the antecubital vein of each participant. The blood samples will be preserved in EDTA tubes and sent to a laboratory for further analysis, including:

Hematological Inflammation Indices: Systemic Immune-Inflammation Index (SII), Aggregate Index of Systemic Inflammation (AISI), Complete blood count with quantitative and percentage analysis, Indicator of Peri-Implantitis and Periodontal Disease Development: morphology by quantitative and percentage separation, Lipid profile: (CHOL , HDL, LDL, TG, APOA1, APOB);

* Inflammatory markers: CRP, ESR, ALB, TP, TF, FIB;
* Cytokine profile: TNF, IL- 1β, IL-6, IL-8, IL-10;
* HOMA2 Parameters: Glucose, Insulin, C-Peptide, HBA1;
* Thyroid profile:- TSH, FT3, FT4, T3, T4, rT3;
* Vitamin D level - 25(OH)D, 1.25(OH)2 D3 Laboratory and Surgical Procedures Each partner institution will conduct laboratory tests and clinical procedures at their respective clinical locations, in collaboration with a certified analytical laboratory.

Next, each participant will undergo implant explantation surgery, during which tissue samples will be collected for further analysis, followed by immediate bone defect regeneration at the implantation site. The procedure will be preceded by removal of the prosthetic restoration.

Following oral disinfection with a 0.2% alcohol-based chlorhexidine solution, local infiltration anesthesia will be administered using 2% articaine with epinephrine 1:200,000. A flap incision will be performed to access the peri-implant region.

A trephine drill with the smallest possible diameter will then be selected to encompass the implant collar. Using the following drilling parameters-800 rpm, 20 Ncm torque, and 0.9% NaCl irrigation-the drill will be lowered to the apical depth of the implant. The implant will be extracted along with any bone tissue tightly adhered to its surface.

The implant and bone tissue will be preserved in a 5% formalin solution. The surgical site will be sutured using non-resorbable 5-0 monofilament sutures.

Both specimens will be sent to research centers in Poland. The implant and tissue samples will be transferred to the Department of Inorganic Chemistry, Analytical Chemistry, and Electrochemistry at the Silesian University of Technology in Gliwice, Poland.

Laboratory Analysis

In the laboratory, biological material will be separated from the samples. The following analyses will be performed:

Titanium concentration measurement and detection of other metals present in the titanium alloy.

Implant surface will be analysed using: Light microscopy, Scanning electron microscopy (SEM), corrosion testing. The microscopic examination will assess the implant surface, identifying areas with fatigue-related material degradation, such as microcracks.

Post-Explantation Follow-Up

One week after the explantation procedure, a follow-up visit will take place. During this visit:

Surgical sutures will be removed. The healing process of the surgical wound will be assessed. If no complications are detected, the next follow-up visit will be scheduled four weeks later. During the four-week follow-up visit, the following evaluations will be performed:

Clinical assessment of the implantation site, including HKT and WKT parameters A second CBCT scan: to assess bone structure in the post-implantation region, with measurements including: Percentage of bone loss, calculated as the ratio of the smallest vertical dimension of the alveolar ridge in the post-implantation area to the height of the alveolar ridge in the immediate vicinity

Blood Sample Collection:

20ml of venous blood will be collected from the antecubital vein of each participant.

The blood sample will be preserved in EDTA tubes and sent to an analytical laboratory for further testing, including same parameters as mentioned previously.

ELIGIBILITY:
Inclusion Criteria:

* PD (Pocket Depth) at the implant site exceeds 6mm,
* Positive BoP (Bleeding on Probing) index
* Bone loss exceeding 66% on at least one implant surface

Exclusion Criteria:

* General and local contraindications for surgical procedures
* Pregnancy
* Use of bisphosphonates or other antiresorptive medications in medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood testing, total blood count, and indices derived from it. | On the day of implant removal (before implant removal) and 4 weeks after.
  Hematological Inflammation Indices: Systemic Immune-Inflammation Index (SII) calculated as follows: SII=NEUxPLT/LYMPH
Blood testing, total blood count, and indices derived from it. | On the day of implant removal (before implant removal) and 4 weeks after.
  Hematological Inflammation Indices: Aggregate Index of Systemic Inflammation (AISI) calculated as follows: AISI= NEU×PLTxMON/LYMP
Blood testing, lipid profile. | On the day of implant removal (before implant removal) and 4 weeks after.
  CHOL mg/dl , HDL mg/dl, LDL mg/dl, TG mg/dl, APOA1 mg/dl, APOB mg/dl
Blood testing, Inflammatory markers. | On the day of implant removal (before implant removal) and 4 weeks after.
  Inflammatory markers: CRP mg/l, albumin (ALB) mg/dl, TP mg/dl,TF mg/dl, FIB mg/dl
Blood testing, Inflammatory marker. | On the day of implant removal (before implant removal) and 4 weeks after.
  ESR mm/h
Blood testing, Cytokine profile. | On the day of implant removal (before implant removal) and 4 weeks after.
  TNF- α pg/ml , IL- 1β pg/ml, IL-6 pg/ml, IL-8 pg/ml, IL-10 pg/ml
Blood testing, HOMA2 Parameters | On the day of implant removal (before implant removal) and 4 weeks after.
  HOMA2 Parameters - Glucose mg/dl, C-Peptide mg/dl,
Blood testing, HOMA2 Parameters | On the day of implant removal (before implant removal) and 4 weeks after.
  Insulin mU/ml
Blood testing, HOMA2 Parameters | On the day of implant removal (before implant removal) and 4 weeks after.
  HBA1C %
Blood testing, Thyroid profile | On the day of implant removal (before implant removal) and 4 weeks after.
  TSH μIU/ml
Blood testing, Thyroid profile | On the day of implant removal (before implant removal) and 4 weeks after.
  FT3 ng/l, FT4 ng/l
Blood testing, Thyroid profile | On the day of implant removal (before implant removal) and 4 weeks after.
  T3 ng/dl, T4 ng/dl
Blood testing, Thyroid profile | On the day of implant removal (before implant removal) and 4 weeks after.
  rT3 ng/ml
Blood testing, Vitamin D3 level | On the day of implant removal (before implant removal) and 4 weeks after.
  25(OH)D, 1.25(OH)2 D3 ng/ml
Clinical examination - general, oral cavity | On the day of implant removal (before implant removal) and 4 weeks after.
  Oral Hygiene Index (OHI) %, Aproximal Plaque Index (API) %
Clinical examination - general, oral cavity, utilizing a UNC15 periodontal probe | On the day of implant removal (before implant removal).
  Community Index of Periodontal Treatment Needs (CPITN)
Clinical examination - implant site, utilizing a UNC15 periodontal probe | On the day of implant removal (before implant removal).
  Pocket Depth (PD) - measured on four surfaces around the implant in mm.
Clinical examination - implant site, utilizing a UNC15 periodontal probe | On the day of implant removal (before implant removal).
  Bleeding on Probing (BoP) Index - Yes or No. (0 or 1).
Clinical examination - implant site, utilizing a UNC15 periodontal probe | On the day of implant removal (before implant removal).
  Width and height of the attached gingiva (HKT, WKT) in mm.
Clinical examination - implant site, utilizing a UNC15 periodontal probe | On the day of implant removal (before implant removal).
  Possible implant mobility, assessed using the Mobility Index (MOB) acc to Misch, Grade: 0,1,2 or 3
Radiology-based evaluation | On the day of implant removal (before implant removal).
  Cone-Beam Computed Tomography: Bone loss percentage on the implant site (%), calculated as the ratio of bone defect depth from the implant platform to the base of the defect, relative to the total implant length, assessed separately for each of the four implant surfaces (mesial, distal, buccal, and lingual/palatal)
Radiology-based evaluation | On the day of implant removal (before implant removal) and 4 weeks after.
  Cone-Beam Computed Tomography: Bone density on the implant site (before and after implant removal), measured in Hounsfield units (HU)
Implant surface evaluation, light microscopy | Within 48 hours after implant removal
  Assessment of the implant surface, identifying areas with fatigue-related material degradation, such as microcracks.
Implant surface evaluation, Scanning electron microscopy | Within 48 hours after implant removal
  Assessment of the implant surface, identifying areas with fatigue-related material degradation, such as microcracks.
Implant surface evaluation - detection of other metals presented in the titanium alloy. | Within 48 hours after implant removal
  Energy-dispersive X-ray spectroscopy (EDS)
Titanium ions concentration in tissues attached to implant' surface | Within 48 hours after implant removal
  Inductively coupled plasma mass spectrometry (ICP-MS)

CONTACTS AND LOCATIONS:
Overall Officials: Marzena Dominiak, Prof, Study Chair — Wroclaw Medical Univeristy
Locations (1):
- Oral Surgery Department Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
All collected anonymized IPD will be available on Zenodo Repository.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 12 months after finishing the study.
Access Criteria: All anonymized (due to General Data Protection Policy) data will be available on demand.
URL: https://zenodo.org/

REFERENCES:
- [Background] Elani HW, Starr JR, Da Silva JD, Gallucci GO. Trends in Dental Implant Use in the U.S., 1999-2016, and Projections to 2026. J Dent Res. 2018 Dec;97(13):1424-1430. doi: 10.1177/0022034518792567. Epub 2018 Aug 3. PMID 30075090
- [Background] Fu JH, Wang HL. Breaking the wave of peri-implantitis. Periodontol 2000. 2020 Oct;84(1):145-160. doi: 10.1111/prd.12335. PMID 32844418
- [Background] Schwarz F, Claus C, Becker K. Correlation between horizontal mucosal thickness and probing depths at healthy and diseased implant sites. Clin Oral Implants Res. 2017 Sep;28(9):1158-1163. doi: 10.1111/clr.12932. Epub 2016 Jul 26. PMID 27458093
- [Background] Schwarz F, Derks J, Monje A, Wang HL. Peri-implantitis. J Periodontol. 2018 Jun;89 Suppl 1:S267-S290. doi: 10.1002/JPER.16-0350. PMID 29926957
- [Background] Albrektsson T, Canullo L, Cochran D, De Bruyn H. "Peri-Implantitis": A Complication of a Foreign Body or a Man-Made "Disease". Facts and Fiction. Clin Implant Dent Relat Res. 2016 Aug;18(4):840-9. doi: 10.1111/cid.12427. Epub 2016 May 30. PMID 27238274
- [Background] Pettersson M, Kelk P, Belibasakis GN, Bylund D, Molin Thoren M, Johansson A. Titanium ions form particles that activate and execute interleukin-1beta release from lipopolysaccharide-primed macrophages. J Periodontal Res. 2017 Feb;52(1):21-32. doi: 10.1111/jre.12364. Epub 2016 Mar 14. PMID 26987886
- [Background] Tsave O, Petanidis S, Kioseoglou E, Yavropoulou MP, Yovos JG, Anestakis D, Tsepa A, Salifoglou A. Role of Vanadium in Cellular and Molecular Immunology: Association with Immune-Related Inflammation and Pharmacotoxicology Mechanisms. Oxid Med Cell Longev. 2016;2016:4013639. doi: 10.1155/2016/4013639. Epub 2016 Apr 11. PMID 27190573
- [Background] Scibior A, Pietrzyk L, Plewa Z, Skiba A. Vanadium: Risks and possible benefits in the light of a comprehensive overview of its pharmacotoxicological mechanisms and multi-applications with a summary of further research trends. J Trace Elem Med Biol. 2020 Sep;61:126508. doi: 10.1016/j.jtemb.2020.126508. Epub 2020 Apr 12. PMID 32305626
- [Background] Grande F, Tucci P. Titanium Dioxide Nanoparticles: a Risk for Human Health? Mini Rev Med Chem. 2016;16(9):762-9. doi: 10.2174/1389557516666160321114341. PMID 26996620
- [Background] Zhang HM, Cao J, Tang BP, Wang YQ. Effect of TiO(2) nanoparticles on the structure and activity of catalase. Chem Biol Interact. 2014 Aug 5;219:168-74. doi: 10.1016/j.cbi.2014.06.005. Epub 2014 Jun 12. PMID 24931876
- [Background] Chen WQ, Zhang SM, Qiu J. Surface analysis and corrosion behavior of pure titanium under fluoride exposure. J Prosthet Dent. 2020 Aug;124(2):239.e1-239.e8. doi: 10.1016/j.prosdent.2020.02.022. Epub 2020 May 10. PMID 32402439
- [Background] Trepanier C, Tabrizian M, Yahia LH, Bilodeau L, Piron DL. Effect of modification of oxide layer on NiTi stent corrosion resistance. J Biomed Mater Res. 1998 Winter;43(4):433-40. doi: 10.1002/(sici)1097-4636(199824)43:43.0.co;2-#. PMID 9855202
- [Background] Chouirfa H, Bouloussa H, Migonney V, Falentin-Daudre C. Review of titanium surface modification techniques and coatings for antibacterial applications. Acta Biomater. 2019 Jan 1;83:37-54. doi: 10.1016/j.actbio.2018.10.036. Epub 2018 Oct 26. PMID 30541702